CLINICAL TRIAL: NCT07356908
Title: Short- Term Outcome and One -Year Recurrence in Acute Pulmonary Embolism Patients With and Without Sleep - Disordered Breathing
Brief Title: Impact of Sleep Related Breathing Disorders on Outcomes of Acute Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Sponsor
Other Study IDs: fac med; faculty of medicin (Other: Alexandria University)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Embolism; Sleep Apnea Syndrome (OSAS)
Keywords: pulmonary embolism; sleep apnea
MeSH Terms: conditions — Pulmonary Embolism; Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: polysomnography — This prospective observational study will include consecutive adult patients admitted to the Chest Diseases Department and related units at Alexandria Main University Hospital (AMUH) with a diagnosis of acute pulmonary embolism confirmed by CTPA

SUMMARY:
This study aimsto compare short-termclinical outcomesand one-year recurrence rates in patients with acute pulmonary embolism with versus without sleep-disordered breathing, recruited from Alexandria MainUniversityHospital.

DETAILED DESCRIPTION:
This prospective observational study will include consecutive adult patients admitted to the Chest Diseases Department and related units at Alexandria Main University Hospital (AMUH) with a diagnosis of acute pulmonary embolism confirmed by CT pulmonary angiography and followed up with sllep study to asses the effect of sleep related breathing disorderon the recurrence of emboli.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18years.

  * Objectively confirmed acute pulmonary embolism by computed tomography pulmonary angiography (CTPA).
  * Hemodynamically stable or clinically stabilized within 72 hours of admission. .Ability to provide informed consent.

Exclusion Criteria:

.Known central sleep apnea without obstructive features. .Inabilityto undergo sleep study evaluation.

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients more than 18 years diagnosed with pulmonary embolism managed and followed up at the chest diseases department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary embolism recurrence | 12 months
  ocuurence of pulmonary embolism during the follow up period confirmed by CTPA
Recurrence of Pulmonary Embolism | ONE YEAR
  occurence of objectively confirmed pulmonary embolism during the one t=year follow up period confirmed by CTPA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
refusal by the department

REFERENCES:
- See also: Alonso-Fernández A, de la Peña M, Romero D, Piérola J, Carrera M, Barceló A, Soriano JB, García Suquia A, Fernández-Capitán C, Lorenzo A, García-Río F. Association between obstructive sleep apnea and pulmonary embolism. Mayo Clin Proc. 2013 Jun;88(6):579 — https://pubmed.ncbi.nlm.nih.gov/23578813/
- Available data/document: Study Protocol: Alonso-Fernández A, de la Peña — https://pubmed.ncbi.nlm.nih.gov/23578813/ — https://pubmed.ncbi.nlm.nih.gov/23578813/.